CLINICAL TRIAL: NCT04443647
Title: Influence of Oxytocin on Approach-avoidance Tendencies to Social and Non-social Stimuli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Prof. dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SingleOT_EEG-App-avoid_S56327
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Basic Science
Keywords: oxytocin; sociality; approach-avoidance motivational tendencies; EEG frontal assymmetry; skin conductance; autonomic arousal
MeSH Terms: conditions — Social Behavior | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Syntocinon nasal spray (40 IU/ml; oxytocin, product code RVG 03716); single intranasal dose of 24 international units (IU; 3 puffs of 4 IU per nostril)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Saline natriumchloride solution nasal spray; single intranasal dose (3 puffs per nostril)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Syntocinon nasal spray
  Arms: Oxytocin
Drug: Placebo — Placebo nasal spray
  Arms: Placebo

SUMMARY:
In this study, a randomized, placebo-controlled between-subject design is adopted to investigate the effect of a single-dose of intranasally administered OT on approach-avoidance related motivational tendencies during the processing of a series of social and non-social, positively and negatively valenced stimuli. To obtain a behavioral measure of approach-avoidance tendencies, participants will be able to control the viewing time of the presented stimuli, by pressing 'up' or 'down' on a keyboard. During stimulus presentation neurophysiological recordings will be performed to obtain a neural measure of approach-avoidance motivational tendencies, based on electroencephalographic recordings (EEG: frontal alpha asymmetry). Also assessments of autonomic arousal, based on skin conductance recordings will be collected.

DETAILED DESCRIPTION:
The neuropeptide oxytocin (OT) plays an important role in a wide-range of complex social behaviors. Recently however, the 'social' specificity of OT's action has been challenged, considering several observations of non-social effects of OT showing for example that OT reliably reduces stress also in non-social tasks.

To account for these non-social effects of OT, the General Approach-Avoidance Hypothesis of OT (GAAO) has been put forward, positing that OT primarily modulates approach/ avoidance motivational tendencies and behaviors by impacting on the mesocorticolimbic circuitry linked to reward (approach) as well as cortico-amygdala circuits linked to threat (avoidance) (Harari-Dahan and Bernstein, 2014). Since the neural substrates underlying 'social' approach and avoidance are not distinct from those underlying 'non-social' approach and avoidance, the GAAO posits that the modulatory effects of OT should not be limited to social behaviors. In this view, the GAAO puts forward that OT may indeed enhance the attentional salience of many social cues, but not because they are social per se; but because many social stimuli are emotionally-evocative and personally-relevant.

In this study, a randomized, placebo-controlled between-subject design is adopted to investigate the effect of a single-dose of intranasally administered OT on approach-avoidance related motivational tendencies during the processing of a series of social and non-social, positively and negatively valenced stimuli. To obtain a behavioral measure of approach-avoidance tendencies, participants will be able to control the viewing time of the presented stimuli, by pressing 'up' or 'down' on a keyboard. During stimulus presentation neurophysiological recordings will be performed to obtain a neural measure of approach-avoidance motivational tendencies, based on electroencephalographic recordings (EEG: frontal alpha asymmetry). Also electrodermal recordings (skin conductance) will be collected to obtain assessments of sympathetically-driven autonomic arousal.

In accordance to the GAAO account, it is hypothesized that OT will reduce avoidance-related motivational tendencies (assessed behaviorally and using EEG), irrespective of sociality (i.e. similar effect towards social and non-social stimuli).

In accordance to prior research, skin conductance responses are hypothesized to reduce after OT, indicating reduced sympathetically-driven autonomic arousal. On the other hand, considering the implicated role of sympathetic arousal in orienting responses, OT might also facilitate an enhancement of skin conductance responses, i.e., being reflective of OT's role in enhancing salience toward emotionally-evocative stimuli.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* male
* age between 18 and 35
* Normal or adjusted-to-normal vision (with lenses only)
* Dutch as mother tongue

Exclusion Criteria:

* female
* age below 18 or above 35
* neurological or psychiatric condition (e.g. epilepsy, stroke, concussion), (e.g. anxiety disorder, depression)
* use of psychotropic medication (e.g. anxiolytics, antidepressants)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in EEG frontal alpha asymmetry after nasal spray administration | Average over trials, baseline and approximately 30 minutes after nasal spray administration
  The influence of oxytocin administration on EEG frontal alpha asymmetry
Change in behavioral approach-avoidance (number of up or down key presses, prolonging or shortening the viewing time towards presented stimuli) | Average over trials, baseline and approximately 30 minutes after nasal spray administration
  During the presentation of a series of stimuli, participants will be able to prolong or shorten the viewing time towards the presented stimuli, by pressing an 'up' or 'down' key on a keyboard. The number of up versus down key-presses will be taken as a measure of behavioral approach-avoidance.
  The influence of oxytocin administration on the number of up or down key presses will be assessed.
Change in skin conductance (type of electrodermal recording) after nasal spray administration | Average over trials, baseline and approximately 30 minutes after nasal spray administration
  The influence of oxytocin adminstration on skin conductance

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data will be made availabe to other researchers upon reasonable request.

REFERENCES:
- [Background] Harari-Dahan O, Bernstein A. A general approach-avoidance hypothesis of oxytocin: accounting for social and non-social effects of oxytocin. Neurosci Biobehav Rev. 2014 Nov;47:506-19. doi: 10.1016/j.neubiorev.2014.10.007. PMID 25454355
- [Derived] Alaerts K, Taillieu A, Daniels N, Soriano JR, Prinsen J. Oxytocin enhances neural approach towards social and non-social stimuli of high personal relevance. Sci Rep. 2021 Dec 8;11(1):23589. doi: 10.1038/s41598-021-02914-8. PMID 34880300